CLINICAL TRIAL: NCT05657561
Title: The Effect of Early Mobilization Training on Mobility, Pain and Comfort After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevinç Taştan, Prof. Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FD_01
Record Dates: First submitted 2022-11-27; First posted 2022-12-20 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Abdominal Surgery
Keywords: abdominal surgery; early mobilization
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: Experimental study with pretest posttest control group
Masking Description: Patients who have had abdominal surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early mobilization (Experimental): Patients in the intervention group will be given "Early Mobilization Training" in the preoperative preparation unit in the preoperative period.
  Interventions: Other: early mobilization
- routine clinical care (No Intervention): Patients in the control group will receive routine clinical care .Routine post-operative mobilization procedure will be delivered by clinic doctors and nurses

INTERVENTIONS:
Other: early mobilization — Mobilization training was given to the intervention group.
  Arms: early mobilization

SUMMARY:
The primary aim of this study is to examine the effects of in-bed rotation and early mobilization training given before abdominal surgery on mobility, pain and comfort of patients after surgery. The secondary aim of the study is to examine the effect of mobilization training given before abdominal surgery on the sleep of patients after surgery.

DETAILED DESCRIPTION:
The primary aim of this clinical trial study is to examine the effects of early mobilization training given before abdominal surgery on mobility, pain and comfort of patients after surgery. The secondary aim of the study is to examine the effect of mobilization training given before abdominal surgery on the sleep of patients after surgery. Research Hypotheses are:

H11. There is a difference between the mobility scores of the patients who were given and not given pre-abdominal surgery training.

H12. There is a difference between the comfort scores of patients who were given and not given pre-abdominal surgery training.

H13. There is a difference between the sleep scores of the patients who were given and not given pre-abdominal surgery training.

First, the patient's mobility status in the preoperative period was evaluated with these scales. "Early Mobilization Training" will be given to the patients in the intervention group in the preoperative period. "Early Mobilization Training Material" to be prepared by the researcher will be used as training material. The training content will include information about the techniques and points to be considered about turning from one side to the other in the bed, sitting on the side of the bed, standing on the side of the bed and walking in the patient's room, and the time spent outside the bed on the day of surgery and the first and subsequent days after surgery.

After the patient's mobilization on the first day after the operation, the Patient Mobility Scale, the Postoperative Mobilization, the Visual Analogue Scale (VAS) questions questioning the pain and comfort during lying and sitting, and sleep status will be filled.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* those with abdominal surgery

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Mobility Scale | Change in Baseline Patient mobility score at two days
  he level of pain and difficulty experienced during the 4 post-surgical activities (turning from one side of the bed to the other, sitting by the bed, standing up at the bedside, and walking in the patient's room) is evaluated using a 15 cm visual analog with verbal expressions listed at the bottom along the scale.
  The numerical value of the degree of pain and difficulty is determined by measuring the distance between the mark on the scale and "0" with a calibrated ruler. An increase in scores indicates an increase in pain and difficulty related to activity. The scores obtained give the patient's mobility score for each activity. The average score value is calculated. Scores for all activities are added together to obtain the global patient mobility score. The total score that can be obtained from the scale varies between 0-120.

SECONDARY OUTCOMES:
pain level | Change in Baseline Patient pain score at two days
  Preoperative and postoperative pain levels of the patients will be measured with the Visual Anolog Scale for pain.The Visual Analog Scale is a self-reported based measurement tool that is often used to measure subjective experiences pain. In this study, Visual Analog Scale for pain was used to make a numerical definition of a participant's pain levels with the participants' self-reports. Numbers between 0-10 were defined on a line, and the participants were asked to indicate the number of pain intensity levels they feel on this line. Participants with no pain scored 0 and extremely pain participants scored 10.
comfort level in bed and while sitting | Change in Baseline comfort score at two days
  The comfort level of the patients while turning and sitting in bed will be measured with the Visual Analog Scale for Comfort. In this study, Visual Analog Scale for comfort was used to make a numerical definition of a participant's comfort levels with the participants' self-reports. Numbers between 0-10 were defined on a line, and the participants were asked to indicate the number of comfort intensity levels they feel on this line. Participants with no comfort scored 0 and extremely comfort participants scored 10.

CONTACTS AND LOCATIONS:
Overall Officials: Sevinc Tastan, Prof., Study Director — Eastern Mediterranean University, Health Sciences Faculty, Famagusta, North Cyprus,
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Shea G. Ventricular assist devices: what intensive care unit nurses need to know about postoperative management. AACN Adv Crit Care. 2012 Jan-Mar;23(1):69-83; quiz 84-5. doi: 10.1097/NCI.0b013e318240aaa9. PMID 22290092
- [Background] Auyong DB, Allen CJ, Pahang JA, Clabeaux JJ, MacDonald KM, Hanson NA. Reduced Length of Hospitalization in Primary Total Knee Arthroplasty Patients Using an Updated Enhanced Recovery After Orthopedic Surgery (ERAS) Pathway. J Arthroplasty. 2015 Oct;30(10):1705-9. doi: 10.1016/j.arth.2015.05.007. Epub 2015 May 12. PMID 26024988
- [Background] Adler J, Malone D. Early mobilization in the intensive care unit: a systematic review. Cardiopulm Phys Ther J. 2012 Mar;23(1):5-13. PMID 22807649
- [Background] Castelino T, Fiore JF Jr, Niculiseanu P, Landry T, Augustin B, Feldman LS. The effect of early mobilization protocols on postoperative outcomes following abdominal and thoracic surgery: A systematic review. Surgery. 2016 Apr;159(4):991-1003. doi: 10.1016/j.surg.2015.11.029. Epub 2016 Jan 21. PMID 26804821
- [Background] Chen LC, Wang TF, Shih YN, Wu LJ. Fifteen-minute music intervention reduces pre-radiotherapy anxiety in oncology patients. Eur J Oncol Nurs. 2013 Aug;17(4):436-41. doi: 10.1016/j.ejon.2012.11.002. Epub 2012 Dec 4. PMID 23218591
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Park DI, Kim HJ, Park JH, Cho YK, Sohn CI, Jeon WK, Kim BI, Ryu SH, Sung IK. Factors affecting abdominal pain during colonoscopy. Eur J Gastroenterol Hepatol. 2007 Aug;19(8):695-9. doi: 10.1097/01.meg.0000219097.32811.24. PMID 17625440
- [Background] Hashem MD, Nelliot A, Needham DM. Early Mobilization and Rehabilitation in the ICU: Moving Back to the Future. Respir Care. 2016 Jul;61(7):971-9. doi: 10.4187/respcare.04741. Epub 2016 Apr 19. PMID 27094396
- See also: Postoperative Pain Control — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3747287/
- See also: Ambulatory care nursing-sensitive indicators — https://journals.lww.com/nursingmanagement/fulltext/2016/06000/ambulatory_care_nursing_sensitive_indicators.7.aspx?casa_token=SSRmATEPZagAAAAA:2ZP0eWy3Ms3-jbtZal1gjR3EVgIM7bKieDbcgSw_hKSopRmkHDuXbsAs30G2Y6isOoPejMZxOrqM5AtF1aMybe4